CLINICAL TRIAL: NCT07320196
Title: The Effectiveness of Smart Mind Maps in Promoting Safe Administration of High-Alert Medications Among Nurses in the Pediatric Intensive Care Unit
Brief Title: Smart Mind Maps in Promoting Safe Administration of High-Alert Medications
Acronym: HAMs- PICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Mind Map high alert medication
Record Dates: First submitted 2025-09-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: PICU; Nurses
Keywords: HAMs; PICU; Nurses; Safe administration

STUDY DESIGN:
Intervention Model Description: The study will include a convenience sample comprising of all nurses available and on duty in the PICU (who directly handled HAM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one group pretest/post test (Experimental): PICU nurses who directly handled HAM
  Interventions: Other: smart mind mapsde

INTERVENTIONS:
Other: smart mind mapsde — designing a smart mind maps as an advanced conceptual tool to help nurses understand well about HAMs

SUMMARY:
In PICU setting, drug administration, monitoring, and prescribing errors made up most cases (54%) of MEs . Emphasizes these issues requires a multifaceted approach, including staff training, creation of innovative cognitive frameworks, use of electronic prescribing systems, and the promotion of a safety-awareness within healthcare settings. Recently, mind mapping has been applied in the field of nursing education as an advanced conceptual tool. It uses a technique of combining drawings with words to build memory associations between a topic keyword and image, color, or other link allowing learners to effectively store and extract information

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of smart mind maps in promoting safe administration of high-alert medications among nurses in the pediatric intensive care unit. Designing a mind map using AI holds significant value for nurses working in the PICU. AI-powered mind maps can help nurses organize complex patient information more efficiently, enabling quicker decision-making and improved care planning. By integrating AI, the mind map can automatically update with real-time data, alert nurses to critical changes, and even suggest evidence-based interventions. This not only enhances patient safety and care quality but also reduces cognitive load and streamlines communication among the healthcare team .

ELIGIBILITY:
Inclusion criteria:

* Nurses on duty in the PICU (who directly handled HAM) irrespectively to their age, sex, educational level.

Exclusion Criteria:

* Nurses who do not handle with HAM

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tool I: A Structured Assessment Questionnaire | 2 weeks
  It will be developed by the researcher which will consist of two parts:
  Part 1: Socio-demographic Characteristics and Professional Data of Studied Nurses part 2: Knowledge Assessment Tool on AI and Mind Mapping for Nurses (pre/posttest)
Tool II: Nurses' Knowledge Regarding Safe Use of High-Alert Medications (HAMs) | 1 month
  It will be developed to collect data necessary for evaluating nurses' knowledge related to safe use of high-alert medications. The assessment will encompass key domains such as the definition and classification of HAMs, safety precautions during drug administration (including delivery routes and dosage accuracy), and drug regulation (including proper storage, documentation, and handling procedures).
Tool III: Observational Checklist for Safe Handling of High Alert Medications | 2 month
  It will be developed by the researcherto objectively assess nurses' practices related to the safe handling of high-alert medications in PICUs according to the international recognized guidelines and evidence-based protocols.

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared because the study involves sensitive clinical data from a small population, and sharing may pose confidentiality risks despite de-identification.
  Access Criteria:
  Not applicable. IPD will not be shared.

REFERENCES:
- See also: Related Info — https://doi.org/10.21608/jnsbu.2023.319643